CLINICAL TRIAL: NCT06275945
Title: Feasibility Study of A VoRo UrologIc ScaffolD for the Prophylactic Treatment of Post-Prostatectomy Stress Urinary Incontinence
Brief Title: Feasibility Study of A VoRo UrologIc ScaffolD (ARID)
Acronym: ARID
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Levee Medical, Inc. (Industry)
Collaborators: RQM+ (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1010073
Record Dates: First submitted 2024-02-08; First posted 2024-02-23 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Stress Urinary Incontinence; Radical Prostatectomy
Keywords: SUI; Radical Prostatectomy
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized first-in-man study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Voro Urologic Scaffold Group (Experimental): Subjects undergo radical prostatectomy procedure as part of their stand of care treatment for their prostate cancer. The Voro Urologic Scaffold is placed during the prostatectomy procedure after prostate removal. The device is placed over the urethral stump in its compressed configuration. With the device compressed at the pelvic floor, the urethral stump is anastomosed with the bladder neck. The device is expanded and positioned over the anastomosed urethra and bladder neck. The distal end of the device is sutured in place and the proximal end of the device is sutured to the bladder.
  The time of Voro Urologic Scaffold insertion and time of completion of device placement (i.e., final sutures placed) will be recorded.
  Incision closure will proceed per institution standard of care for the radical prostatectomy procedure.
  Interventions: Device: Voro Urologic Scaffold

INTERVENTIONS:
Device: Voro Urologic Scaffold — radical prostatectomy

SUMMARY:
The objective of this study is to evaluate the safety and performance of the Voro Urologic Scaffold as a prophylactic treatment for post-prostatectomy stress urinary incontinence.

The study is a prospective, multicenter, single arm study. Up to 40 subjects will be treated at up to 3 investigational sites in Panama. Subjects will be followed up post-treatment at catheter removal, 6 weeks post prostatectomy, 3 months, 6 months, 12 months and 2 years.

DETAILED DESCRIPTION:
Approximately 300,000 men undergo radical prostatectomy (RP) worldwide for the treatment of prostate cancer. RP has favorable oncology outcomes but carries risks of erectile dysfunction and urinary incontinence. Urinary incontinence after RP has negatively affects patient quality of life.

The bioresorbable Voro Urologic Scaffold is designed to be placed over the anastomotic site during an RP procedure, between the bladder neck and urethral stump, to constrain the urethra immediately proximal to the urinary sphincter. The device is designed to relieve the load on the urinary sphincter. As the anastomosis heals, connective tissues form in the scaffold geometry while the scaffold material resorbs and hence potentially reduce the risk of acute and chronic stress incontinence.

The objective of this study is to evaluate the safety and performance of the Voro Urologic Scaffold as a prophylactic treatment for post-prostatectomy stress urinary incontinence.

The study is a prospective, multicenter, single arm study. Up to 40 subjects will be treated at up to 3 investigational sites in Panama. Subjects will be followed up post-treatment at catheter removal, 6 weeks post prostatectomy, 3 months, 6 months, 12 months and 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male 45-70 years of age
2. Diagnosed with prostate cancer and scheduled for radical prostatectomy
3. Gleason Grade Group 3 or lower
4. Prostate size less than 80 grams
5. Able and willing to provide written consent to participate in the study
6. Able and willing to comply with study follow-up visits and procedures

Exclusion Criteria:

1. Malignant tumors outside of the prostate capsule confirmed via baseline assessments (e.g., mpMRI, bone scan)
2. History of urinary incontinence, including stress or urge urinary incontinence
3. On medications to treat overactive bladder (OAB)
4. Post void residual >200 ml or > 25% voiding volume
5. Presence of urethral stricture or bladder neck contracture
6. Current or chronic urinary tract infection
7. Prior urologic outlet surgical or minimally invasive procedure (e.g., TURP, HoLEP, Rezum, etc.).
8. Prior pelvic radiation or anticipated need for radiation after radical prostatectomy
9. Presence of stones in the bladder
10. History of neurogenic bladder, sphincter abnormalities, or poor detrusor muscle function
11. Body mass index >35
12. Insulin-dependent diabetes mellitus
13. Current uncontrolled diabetes (i.e., hemoglobin A1c ≥7.5%)
14. Intravesical prostatic protrusion (IPP) >5mm
15. History of immunosuppressive conditions (e.g., AIDS, post-transplant)
16. Any significant medical history that would pose an unreasonable risk or make the subject unsuitable for the study per investigator discretion
17. Any cognitive or psychiatric condition that interferes with or precludes direct and accurate communication with the study investigator regarding the study or affect the ability to complete the study quality of life questionnaires
18. Subject currently participating in other investigational studies unless approved by the Sponsor in writing

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
The change in pad weight of 24-hour pad weight test from baseline to post procedure 6-month and 12-month follow-ups. | Baseline, Foley removal (about 2-week post procedure), 6-week, and 3-, 6-, 12- & 24-months follow-ups.
  The pads are pre-weighed prior to providing them to subjects. The test should be started with an empty bladder. The subject will wear pads and perform their normal daily activities for 24 hours.

SECONDARY OUTCOMES:
The change in pad weight of 1-hour pad weight test from baseline to post procedure 6-month and 12-month follow-ups. | Baseline, post-procedure 6-week, and 3-, 6-, 12- & 24-months follow-ups.
  The 1-hour pad test follows a standard protocol. Prior to the 1-hour test, the subject is asked to ensure he is adequately hydrated. This will be determined by the color of the urine during the voiding prior to the start of the test. The urine must be clear or light yellow in color to start the test. If the urine is dark yellow, the subject should be given fluids to drink until the urine is light yellow or close to colorless (proper hydration).
  If voiding is urgent and unavoidable, the test is terminated. Collect voiding volume and repeat the test after re-hydration.
The changes in the standing cough test (SCT) from baseline to post procedure 6-month and 12-month follow-ups. | Baseline, post-procedure 6-week, and 3-, 6-, 12- & 24-months follow-ups.
  The subject must verbally confirm that they have not voided for at least 60 minutes prior to the examination. Examination of the urethral meatus is performed while the subject performs four forceful coughs. Towels or pads are held several inches from the meatus during coughs to collect any urinary leakage. Leakage is evaluated using the Male Stress Incontinence Grading Scale (MSIGS).

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Choi, Study Chair — Founder and CTO, Levee Medical, Inc
Locations (1):
- National Hospital, Panama City, Punta Pacifica, Panama

REFERENCES:
- [Derived] Gahan JC, Espino G, Young M, Bodden E, Ferrandino MN. Initial results with an absorbable urologic scaffold to mitigate early urinary incontinence following radical prostatectomy: the ARID study. World J Urol. 2026 Jan 17;44(1):106. doi: 10.1007/s00345-026-06186-7. PMID 41546699